CLINICAL TRIAL: NCT02687204
Title: Optimization of Enoxaparin Prophylaxis Using Real-time Anti-Factor Xa Levels in Major Reconstructive Surgery Patients
Brief Title: Twice Daily Enoxaparin Prophylaxis in Reconstructive Surgery Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher Pannucci, Assistant Professor, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 86052
Record Dates: First submitted 2016-02-03; First posted 2016-02-22 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Venous Thromboembolism; Deep Venous Thrombosis; Pulmonary Embolus
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enoxaparin prophylaxis (Active Comparator): All enrolled patients will receive twice daily enoxaparin prophylaxis. Patients with identified out of range peak anti-Xa levels will receive real time dose adjustment and will be considered as the experimental arm.
  Interventions: Drug: Twice daily enoxaparin prophylaxis
- Real time dose adjustment (Experimental): Patients with identified out of range peak anti-Xa levels will receive real time enoxaparin dose adjustment
  Interventions: Drug: Real time dose adjustment

INTERVENTIONS:
Drug: Twice daily enoxaparin prophylaxis — Patients will have peak and trough steady state anti-Xa levels drawn. For patients with out of range peak levels, real time enoxaparin dose adjustment using a clinical protocol will be performed. Repeat steady state levels will be checked.
  Other Names: Lovenox
  Arms: Enoxaparin prophylaxis
Drug: Real time dose adjustment — Patients will have peak and trough steady state anti-Xa levels drawn. For patients with out of range peak levels, real time enoxaparin dose adjustment using a clinical protocol will be performed. Repeat steady state levels will be checked.
  Other Names: Lovenox
  Arms: Real time dose adjustment

SUMMARY:
Blood clots that form in the extremities (deep venous thrombosis) and lungs (pulmonary embolus) are feared complications of reconstructive surgery. One in ten patients with symptomatic pulmonary embolus will be dead in 60 minutes. Patients with deep venous thrombosis can develop the post-thrombotic syndrome, known to be a major driver of poor quality of life. These phenomena, broadly known as venous thromboembolism (VTE), have substantial downstream ramifications, and the US Surgeon General and the American Society of Plastic Surgeons (ASPS), among others, have underscored the importance of VTE prevention in surgical patients. Reconstructive surgery, most commonly performed to fix traumatic injuries or defects after cancer excision, often involves borrowing tissue from adjacent or distant areas on the body; reconstructive surgery patients can routinely have surgical injury involving 20% or more of their total body surface area. Injury and resultant inflammation are known to increase metabolism of certain drugs, including those used to prevent VTE after surgery.

Enoxaparin is a blood-thinning medication that decreases likelihood of blood clot formation. Previous research has shown that reconstructive surgery patients who are given enoxaparin after surgery are less likely to develop VTE. However, despite receiving of a standard dose of enoxaparin, many patients still develop this life-threatening complication. The investigators believe that patients metabolize enoxaparin differently based on the degree of surgical injury created during reconstruction, and seek to critically examine enoxaparin metabolism in reconstructive surgery patients. The proposed research will evaluate how enoxaparin affects the blood based on standard, ASPS-recommended dosing after reconstructive surgeries; the investigators will also examine whether the extent of surgical injury alters metabolism as well. Enoxaparin effectiveness will be tracked using anti-Factor Xa (aFXa) levels. If subtherapeutic aFXa levels are observed, the study will also design, implement and test a clinical enoxaparin dose-adjustment protocol to achieve appropriate post-operative aFXa levels. Further research based on these data will examine reduction in VTE risk when aFXa-driven enoxaparin dosing is used.

DETAILED DESCRIPTION:
The ultimate goal of the investigators research is to better understand the interplay between enoxaparin dosing, degree of surgical injury, and blood clots after major reconstructive surgery. Ultimately, this research will expand medicine's understanding of why post-operative VTE occurs, will allow the investigators to individualize a patient's VTE prophylaxis strategy based on their unique characteristics, and will further improve patient safety after reconstructive surgery.

ELIGIBILITY:
Inclusion criteria:

* Adult patients having plastic and reconstructive surgery who are placed on twice daily enoxaparin prophylaxis after surgery.

Exclusion criteria:

* Contraindication to use of enoxaparin.
* Intracranial bleeding/stroke, hematoma or bleeding disorder.
* Known heparin-induced thrombocytopenia
* Creatinine clearance ≤30mL/min
* Serum creatinine >1.6mg/dL
* Epidural anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with a 90-day VTE (either a 90-day DVT or 90-day PE) | 90 days
  Outcome measure number one will be deep venous thrombosis or pulmonary embolus confirmed with imaging within 90 days of the initial surgery.

SECONDARY OUTCOMES:
Number of patients with a 90-day re-operative hematoma | 90 days
  Outcome number two will be bleeding (hematoma) requiring return to the operating room within 90 days of the initial operation.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Pannucci, MD MS, Principal Investigator — University of Utah
Locations (1):
- University of Utah Hospitals, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared.
Supporting Information: SAP
Time Frame: 9/4/18
Access Criteria: American Society of Plastic Surgeons

REFERENCES:
- [Derived] Pannucci CJ, Fleming KI, Agarwal J, Rockwell WB, Prazak AM, Momeni A. The Impact of Once- versus Twice-Daily Enoxaparin Prophylaxis on Risk for Venous Thromboembolism and Clinically Relevant Bleeding. Plast Reconstr Surg. 2018 Jul;142(1):239-249. doi: 10.1097/PRS.0000000000004517. PMID 29649055
- [Derived] Pannucci CJ, Fleming KI, Momeni A, Prazak AM, Agarwal J, Rockwell WB. Twice-Daily Enoxaparin among Plastic Surgery Inpatients: An Examination of Pharmacodynamics, 90-Day Venous Thromboembolism, and 90-Day Bleeding. Plast Reconstr Surg. 2018 Jun;141(6):1580-1590. doi: 10.1097/PRS.0000000000004379. PMID 29608533
- [Derived] Pannucci CJ, Fleming KI. Comparison of face-to-face interaction and the electronic medical record for venous thromboembolism risk stratification using the 2005 Caprini score. J Vasc Surg Venous Lymphat Disord. 2018 May;6(3):304-311. doi: 10.1016/j.jvsv.2017.10.016. Epub 2018 Feb 13. PMID 29452956